CLINICAL TRIAL: NCT06798402
Title: Effectiveness of Ciprofloxacin Intralesional Injection in the Treatment of Cutaneous Leishmaniasis Compared to Sodium Stibogluconate: a Parallel Groups Comparative Trial
Brief Title: Ciprofloxacin Intralesional Injection for the Treatment of Cutaneous Leishmaniasis Compared to Sodium Stibogluconate
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Mustafa University College (Other)
Collaborators: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Hayder Adnan Fawzi, Ass Prof, Al-Mustafa University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALM25-002; apporval no (58) (Other: Research Ethical Approval of Mustansiriyah University/ College of Pharmacy)
Record Dates: First submitted 2025-01-17; First posted 2025-01-29 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Ciprofloxacin; Antimony Sodium Gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intralesional ciprofloxacin (Experimental): Intralesional ciprofloxacin (2 mg/ml, 100 ml, Ciproxin®, Bayer Schering pharma AG, Germany), each lesion was injected based on lesion size (2 mg/cm2). The infiltration of intralesional dose was given once weekly for up to 6 weeks. Treatment will be stopped in patients cured before 6 weeks of treatment, and patients were only asked to come for lesion assessment. A fine insulin needle was used to infiltrate the lesion.
  The lesion was thoroughly infiltrated with the drug solution until the base was completely blanched. Depending on the lesion size, the amount of solution required ranged from 0.2 to 4.0 ml per lesion. No local anesthesia was added. The solutions were injected intralesionally and not subcutaneously.
  Interventions: Drug: Ciprofloxacin (BAYO9867)
- intralesional sodium stibogluconate (Active Comparator): Intralesional sodium stibogluconate (100 mg/ml, 100 ml vial, Pentostam®, GlaxoSmithKline, UK), each lesion was injected based on lesion size (1 mg/cm2).
  The infiltration of intralesional dose was given once weekly for up to 6 weeks. Treatment will be stopped in patients cured before 6 weeks of treatment, and patients were only asked to come for lesion assessment. A fine insulin needle was used to infiltrate the lesion.
  The lesion was thoroughly infiltrated with the drug solution until the base was completely blanched. Depending on the lesion size, the amount of solution required ranged from 0.2 to 4.0 ml per lesion. No local anesthesia was added. The solutions were injected intralesionally and not subcutaneously.
  Interventions: Drug: sodium stibogluconate (Pentostam)

INTERVENTIONS:
Drug: Ciprofloxacin (BAYO9867) — Intralesional ciprofloxacin (2 mg/ml, 100 ml, Ciproxin®, Bayer Schering pharma AG, Germany), each lesion was injected based on lesion size (2 mg/cm2).
  Arms: intralesional ciprofloxacin
Drug: sodium stibogluconate (Pentostam) — Intralesional sodium stibogluconate (100 mg/ml, 100 ml vial, Pentostam®, GlaxoSmithKline, UK), each lesion was injected based on lesion size (1 mg/cm2)
  Arms: intralesional sodium stibogluconate

SUMMARY:
The Aim of the trial to evaluate the effectiveness of intralesional ciprofloxacin 0.2% solution as a local injection in treating cutaneous leishmaniasis and compare its effect with intralesional sodium stibogluconate (SSG) 10% intravenous solution in cutaneous leishmaniasis as a local injection.

In a randomized parallel groups clinical trial, patients were divided into two groups based on therapeutic regimen: 1) intralesional sodium stibogluconate weekly injection and 2) intralesional ciprofloxacin injection. Each lesion was considered a case in the final analysis. Each lesion will be followed up for 90 days (censor endpoint) or until the lesions are cured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single or multiple (less than seven lesions) lesions of cutaneous leishmaniasis

Exclusion Criteria:

* Patients who received anti-leishmaniasis treatment locally or systemically for the last month before this study
* patients on prolonged corticosteroid therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate | From enrollment to the end of treatment up to 90 days.
  Patients were followed weekly up to 90 days after the first injection; four parameters were used for assessment as follows according to Sharquie modified leishmania score:
  1. Measure the size of the lesion through the surface area
  2. Measurement of the induration of the lesion
  3. Assess the degree of erythema of the lesion
  4. Assess the presence and absence of ulceration The obtained data is converted from numbers into scores. The total score was calculated by adding individual scores.
  Score 13-16: Mild response. Score 9-12: Moderate response. Score 5-8: Marked response. Score 0-4: Complete response & clearance Both marked and complete responses are considered as a cure

CONTACTS AND LOCATIONS:
Locations (1):
- Mustansiriyah University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided